CLINICAL TRIAL: NCT07052214
Title: A Single Arm, Multicenter, Prospective, Open Label, Longitudinal Phase 3 Study of Prostate Specific Membrane Antigen (PSMA) Positron Emission Tomography (PET) Combined With Magnetic Resonance Imaging (MRI) Compared to Standard of Care (SOC) for the Detection of Prostate Cancer (PCa).
Brief Title: PSMA PET Combined With MRI for the Detection of PCa
Acronym: BiPASS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Collaborators: Telix Innovations S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-TLX007-CDx-301
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: PCA; Prostate Cancer; Prostatic Neoplasm; PSMA PET; Diagnostic Imaging; Elevated PSA; Positron Emission Tomography; Prostate Biopsy; Carcinoma of the Prostate
Keywords: Molecular Imaging; Biopsy Naive; Magnetic Resonance Imaging; Biopsy; Targeted Biopsy; Radiopharmaceuticals; Cancer Detection; Urologic Oncology
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Illuccix: 68Ga-PSMA-11/Gallium Ga 68 Gozetotide (Other): This is a single arm study. All participants will first undergo mpMRI and PSMA PET scans (one single IV bolus of Gallium Ga 68 Gozetotide administered)
  Interventions: Drug: 68Ga-PSMA-11

INTERVENTIONS:
Drug: 68Ga-PSMA-11 — The radioconjugate 68Ga-PSMA-11 is composed of a human PSMA-targeting ligand peptide conjugated via the acyclic radiometal chelator, N, N'-bis [2-hydroxy-5-(carboxyethyl)benzyl] ethylenediamine-N, N'-diacetic acid (HBED-CC) to the radioisotope Gallium68 ( 68Ga); which binds to PSMA on the surface of cells expressing PSMA, including malignant prostate cancer cells, which usually overexpress PSMA. 68Ga is a β+ (beta) ray emitting radionuclide that allows precise imaging via PET.
  Other Names: Illuccix; Gallium Ga 68 Gozetotide

SUMMARY:
This is an open label, longitudinal Phase 3 study of prostate specific membrane antigen (PSMA) positron emission tomography (PET) combined with magnetic resonance imaging (MRI) compared to standard of care (SOC) for the detection of prostate cancer (PCa).

DETAILED DESCRIPTION:
This is a single arm, multicenter, prospective, open label Phase 3 study with PSMA PET for the detection of PCa. A total of 204 participants will be enrolled from approximately 25 investigative sites in the United States and Australia.

Participants with a clinical suspicion of PCa, who will undergo template biopsy, based on initial MRI (PI-RADs 3-4) within 3 months (92 days) before enrollment and/or based on clinical suspicion (for PI-RADs 1-2) and who have never undergone a prostate biopsy will be eligible for the study. All participants will first undergo MRI and PSMA PET scans, followed by standard 12 core anatomical (2 core six sectors) template biopsy. If the patient does not have a biopsy, their enrollment in the study will be terminated. If additional lesions are detected on MRI and/or PSMA PET, MRI and/or PMSA PET targeted biopsy can be performed (according to clinician judgment).

Both MRI and/or PSMA targeted biopsies will be performed with 2 cores per lesion or as per institutional standards. Clinicians may use PSMA PET to rule out the need for biopsy, in which case, the patient will not have a histopathological SOT and will terminate their enrollment. All biopsy and clinical care decisions are at the discretion of the investigator/clinician (i.e. the clinician may decide to: not biopsy, solely template biopsy, additional targeted biopsies, etc.) Participants presenting with csPCa will undergo therapy/management as per institutional standard, or according to clinician judgment.

Follow-up data will be collected for up to 6-months for select participants (participants with no baseline imaging or histopathological evidence of PCa). Additional imaging, template and/or targeted biopsies may be performed during the follow-up period, at the discretion of the investigator. Any additional biopsy, imaging, clinical, histological, genetic, and intervention data will contribute to the determination of the CSOT. Follow-up will provide longitudinal surveillance to ensure that participants initially evaluated as negative for PCa on both imaging and histopathology are reliably negative.

ELIGIBILITY:
Inclusion Criteria:

1. Male, at least 18 years old.
2. Have a clinical suspicion of PCa, and will undergo template biopsy, based on either: an initial MRI examination (PI-RADS 3-4) within 3 months (92 days) before enrollment, or no MRI evidence (PI-RADs 1-2) within 3 months (92 days) before enrollment, but a clinician indicated intent to proceed with template biopsy due to non-imaging risk factors.

These are non-imaging risk factors that would lead a patient to be considered for a template biopsy (including but not exclusive to):

1. Persistently elevated or rising PSA i. PSA ≥ 3.0 ng/mL ii. Rising PSA velocity (e.g., >0.35-0.75 ng/mL/year over 2-3 years) is also considered suspicious, especially in men with PSA<10ng/mL.
2. High PSA density (PSAD) i. PSA density > 0.15 ng/mL/cm³ is considered high-risk for csPCa. ii. Calculated as PSA (ng/mL) divided by prostate volume (from MRI).
3. Abnormal digital rectal examination (DRE) i. abnormal findings include:

   1. Nodules
   2. Induration
   3. Asymmetry
   4. Fixation of the prostate ii. An abnormal DRE in any PSA range (including <3 ng/mL) increases cancer suspicion.

b) Strong family history of prostate cancer: i. First-degree relative (father or brother) with PCa ii. Any relative diagnosed at <65 years of age iii. Multiple affected relatives iv. Known hereditary cancer syndromes (e.g., BReast CAncer gene [BRCA]1/2, Homeobox protein Hox-B13 [HOXB13] mutations) c) Other high-risk biomarkers i. 4Kscore: ≥ 7.5-10% risk of high-grade PCa ii. PHI (Prostate Health Index): ≥ 35 suggests elevated risk iii. Prostate Cancer Antigen 3 (PCA3) Score: ≥ 35 considered positive and associated with increased risk of PCa.

iv. Any other established biomarker with values in the high-risk range d) Clinical presentation i. Symptoms suggestive of locally advanced disease (e.g., urinary obstruction, bone pain) ii. Prior negative MRI with ongoing clinical concern 3. Prostate biopsy naïve participants. 4. Eastern Cooperative Oncology Group performance status (ECOG PS) ≤2 per FDA guidelines. 5. Have the capacity to understand the study and be able and willing to comply with all protocol requirements. 6. Provides consent for anatomical template with/without targeted biopsy based on clinical risk, MRI and PSMA PET result. 7. Participants must comply with the radiation protection rules (including hospital admissions and isolation) that are used by the treating institution to protect their contacts and the general public, especially if a female partner of the participant is or could be pregnant.

8. Must agree to practice adequate precautions to prevent pregnancy in a female partner and to avoid potential problems associated with radiation exposure to the unborn child (Recommendations related to contraception and pregnancy testing in clinical trials Version 1.1, (CTFG [Clinical Trial Facilitation Group], 2020). Details of contraceptive measures to be taken by male participants and their female partners are described in Appendix 4 of the Protocol.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Has had prior treatment for PCa or prior diagnosis of csPCa.
2. Obvious metastatic disease on prior conventional imaging.
3. Previous diagnosis of cancer of any primary origin (excluding basal cell carcinoma or squamous cell carcinoma of the skin that has undergone potentially curative therapy).
4. Active prostate infection, or urinary test results suggestive of an active urinary tract infection, evident on medical history, within 4 weeks of enrollment.
5. Prior pelvic irradiation
6. Demonstrate radiographic findings of PI-RADS 5.
7. Has abnormalities in physical examination and protocol-specified clinical laboratory tests during the Screening Period that, in the judgment of the investigator, could affect safety or compliance; and/or is deemed not suitable for participating in this trial in the opinion of the investigator.
8. Unable to understand or is unwilling to sign a written informed consent document or to follow investigational procedures in the opinion of the investigator.
9. Is unable to attain or remain in a supine position while a PET/CT scan is being performed or unable to tolerate a PET/CT scan
10. Unable or unwilling to undergo clinical prostate biopsy, has known allergies, hypersensitivity, or intolerance to the investigational drug/comparator or its excipients.
11. Have prior use of radionuclides with an interval of less than 10 effective half-lives before the administration of 68Ga-PSMA-11.
12. Is participating or plans to participate in any experimental drug or device trial during the study period that are considered outside of therapeutic SOC. Studies involving modifications of sequencing or timing of therapeutic regimens/interventions would be deemed eligible to enroll

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate Cancer is for Males only
Enrollment: 204 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months
  To evaluate the diagnostic performance of combined 68Ga-PSMA-11 PET and MRI targeted biopsy for the detection of PCa, using histopathological confirmation as the SOT.
Co-Primary Endpoint | 12 months
  To assess the sensitivity and specificity of 68Ga-PSMA-11 PET as adjunct to MRI or the detection of PCa, confirmed by predefined standard of truth (SOT).

CONTACTS AND LOCATIONS:
Locations (1):
- Australian Prostate Centre, Melbourne N., Victoria, Australia